CLINICAL TRIAL: NCT07100119
Title: A Multiple Ascending Dose Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intrathecally Administered LY4256984 in Participants With Sporadic Amyotrophic Lateral Sclerosis
Brief Title: A Study of LY4256984 in Participants With Sporadic Amyotrophic Lateral Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27427; J6I-MC-OWAA (Other: Eli Lilly and Company); 2025-521295-6 (Other: EU CTR #); U1111-1321-6118 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-07-31; First posted 2025-08-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY4256984 (Cohorts 1-4) (Experimental): Multiple ascending doses (MAD) of LY4256984 administered intrathecally (IT)
  Interventions: Drug: LY4256984
- Placebo (Placebo Comparator): Administered IT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4256984 — Administered IT
  Arms: LY4256984 (Cohorts 1-4)
Drug: Placebo — Administered IT
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how well LY4256984 is tolerated and what side effects may occur in participants with sporadic amyotrophic lateral sclerosis (ALS). The study drug will be administered intrathecally (IT) into the spine. Blood tests will be performed to check how much LY4256984 gets into the bloodstream and how long it takes the body to eliminate it.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite, possible, or probable diagnosis of sporadic amyotrophic lateral sclerosis (ALS) made by a physician experienced with the management of ALS
* ALS symptom onset as determined by the Investigator within 24 months of Screening
* Have a body mass index (BMI) within the range of greater than or equal to 18.0 and less than or equal to 35.0 kilogram per square meter (kg/m²) (inclusive)

Exclusion Criteria:

* Have a history or presence of medical illness including, but not limited to, any cardiovascular, renal, hepatic, gastrointestinal, respiratory, hematological, endocrine, psychiatric, or neurological disease, convulsions, or any clinically significant laboratory abnormality
* Have a history of another neurodegenerative disease or significant dementia/severe cognitive problems
* Have serum alanine aminotransferase (ALT), aspartate transferase (AST), or total bilirubin levels greater than 2 x upper limit of normal.
* Have a significant renal impairment (estimated glomerular filtration rate <60 milliliters per minute [mL/min]/1.73 m²).
* Have a 12-lead electrocardiogram (ECG) abnormality at screening, in the opinion of the investigator, that increases the risks associated with participating in the study
* Show clinically significant abnormalities in lumbar spine previously known or determined by screening lumbar X-ray or fluoroscopy (if performed)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs), Serious Adverse Event(s) (SAEs), and Adverse Event(s) (AEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Approximately Day 253
  A summary of TEAEs, SAEs, and AEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Plasma Area Under the Concentration Versus Time Curve (AUC) of LY4256984 | Baseline up to Approximately Day 253
  PK: Plasma AUC of LY4256984
PK: Plasma Maximum Concentration (Cmax) of LY4256984 | Baseline up to Approximately Day 253
  PK: Plasma Cmax of LY4256984
PK: Cerebrospinal Fluid Concentrations (CSF) of LY4256984 | Baseline up to Approximately Day 253
  PK: CSF Concentrations of LY4256984

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- UZ Leuven, Leuven, Belgium
- Canada (5):
  - Heritage Medical Research Clinic, Calgary
  - Walter Mackenzie Health Sciences Centre, Edmonton
  - London Health Sciences Centre, London
  - Montreal Neurological Institute and Hospital, Montreal
  - Sunnybrook Research Institute, Toronto
- Germany (3):
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin Rostock Sektion für Translationale Neurodegeneration "Albrecht Kossel" Klinik und Poliklinik für Neurologie, Rostock
  - Universitätsklinikum Ulm, Ulm
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Spain (2):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No